CLINICAL TRIAL: NCT00945048
Title: Non-Invasive Determination of Cardiac Output by Electrical Velocimetry Compared With Magnetic Resonance Tomography and Inert Gas Rebreathing Method
Brief Title: Non-Invasive Determination of Cardiac Output by Electrical Velocimetry
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2009-MA
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: electrical velocimetry — determination of cardiac output by electrical velocimetry
Device: inert gas rebreathing — determination of cardiac output by inert gas rebreathing
Device: spirometry — spirometry for testing the ventilatory function
Device: cardiac magnetic resonance imaging (CMR) — CMR examination which delivers the hemodynamic reference parameters

SUMMARY:
The cardiac output (CO) is an important parameter in the diagnosis and therapy of cardiac diseases. The current standard methods for the determination of the CO, however, are either invasive (e.g. right heart catheterization) or technically expendable and expensive (magnetic resonance tomography, MRT). Therefore the aim of the study at hand was to evaluate the electrical velocimetry technique as a new method for determining the CO and to compare this new technique with the Inert Gas Rebreathing Method and with the Magnetic Resonance Tomography

ELIGIBILITY:
Inclusion Criteria:

* Indication for CMR
* Ability of following instructions for electrical velocimetry test, rebreathing test and spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with indication for CMR
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Saur, Dr., Study Director — 1st Department of Medicine; Jens Kaden, Dr., Study Chair — 1st Department of Medicine
Locations (1):
- 1st Department of Medicine, University Hospital Mannheim, Mannheim, Baden-Wurttemberg, Germany